CLINICAL TRIAL: NCT06659627
Title: Fatigue Improvement Through Aerobic Exercise and Cognitive Behavioural Therapy in Patients With Myasthenia Gravis
Brief Title: Interventions Against Fatigue in Patients With Myasthenia Gravis
Acronym: FIT to ACT-MG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Martijn R. Tannemaat, MD PhD, Principal investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL85072.058.23
Record Dates: First submitted 2024-10-15; First posted 2024-10-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Myasthenia Gravis; Fatigue
Keywords: Myasthenia Gravis; Fatigue; Aerobic Exercise Therapy; Cognitive Behavioural Therapy
MeSH Terms: conditions — Myasthenia Gravis; Fatigue | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Three intervention groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers are blinded. After 32 weeks of the last patient the researchers will be unblinded and the study will proceed as an open-label extension study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise therapy (Other): AET will consist of three weekly sessions of aerobic workouts on a bicycle ergometer for a period of 16 weeks. The first training session will be supervised by an experienced physical therapist at the LUMC. Subsequently, participants will perform the remaining workouts at home. One session per week will be carried out independently at home. The other two sessions will be digitally supervised via a digital connection by students, who will be trained and supervised by an experienced physical therapist. During the intervention, training intensity will be adjusted based on the participant's rate of perceived exertion (Borg Rating of Perceived Exertion (RPE) scale).
  Interventions: Behavioral: Aerobic exercise therapy
- Cognitive behavioural therapy (Other): The entire CBT program will be followed digitally through an online platform and will span 12-16 weeks. The program will be tailored to the individual participants' needs and preferences. Every week or every two weeks, the psychologist provides feedback on the finished sessions and gives new assignments. If necessary, the psychologist will contact a participant by phone for additional support.
  Interventions: Behavioral: Cognitive behavioural therapy
- Usual care (Other): Participants are not restricted in their activities, but will be instructed not to start a new exercise or cognitive behavioural program. Chronic physical therapy and psychological counselling in the context of usual care are allowed to continue.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Aerobic exercise therapy — Participants will follow an aerobic exercise therapy program for 16 weeks.
  Arms: Aerobic exercise therapy
Behavioral: Cognitive behavioural therapy — Participants will follow an cognitive behavioural therapy program for 12-16 weeks.
  Arms: Cognitive behavioural therapy
Other: Usual care — Participants do not follow a program, but continue with care as usual
  Arms: Usual care

SUMMARY:
A prospective assessor-blinded randomized clinical trial investigating the effect of aerobic exercise therapy or cognitive behavioural therapy on fatigue in patients with myasthenia gravis.

DETAILED DESCRIPTION:
This study will be a prospective assessor-blinded randomized controlled trial comparing AET and CBT with usual care (UC). For an individual participant, the overall study duration will be 52 weeks with a total intervention duration of 16 weeks. After 32 and 52 weeks the investigators will analyse the data from the activity tracker and approach each participant to digitally complete a total of three questionnaires. After 32 weeks the researchers will be unblinded and the study will proceed as an open-label extension study.

After signing the informed consent form, an activity tracker (Withings Pulse HR) will be provided to all participants. After a four week observation period to evaluate the baseline levels of daily activity, participants will visit the LUMC for baseline measurements and a blood test. After obtaining these baseline characteristics, all participants will be randomly assigned to either AET, CBT or UC.

Participants in the AET group start with an intake meeting with a physical therapist. AET will consist of three weekly sessions of aerobic workouts on a bicycle ergometer for a period of 16 weeks. The first training session will be supervised by an experienced physical therapist at the LUMC. Subsequently, participants will perform the remaining workouts at home. One session per week will be carried out independently at home. The other two sessions will be digitally supervised via a digital connection by students, who will be trained and supervised by an experienced physical therapist. During the intervention, training intensity will be adjusted based on the participant's rate of perceived exertion (Borg Rating of Perceived Exertion (RPE) scale). During each session, the participant is also able to adjust the wattage of that specific training. Training activity and execution will be monitored remotely using the bicycle ergometer and the activity tracker. Adherence and reasons for possible non-adherence will be monitored by the students. Outcome measures will be collected on follow-up immediately after the 16-week intervention.

Participants in the CBT group start with an online intake meeting with a psychologist. The entire CBT program will be followed digitally through an online platform and will span 12-16 weeks. The program will be tailored to the individual participants' needs and preferences. Every week or every two weeks, the psychologist provides feedback on the finished sessions and gives new assignments. If necessary, the psychologist will contact a participant by phone for additional support. Outcome measures will be collected on follow-up immediately after the 16-week intervention.

The outcome measures of the participants in the UC group are obtained after the four week observation period and after 20 weeks follow-up. Participants are not restricted in their activities, but will be instructed not to start a new exercise or cognitive behavioural program. Chronic physical therapy and psychological counselling in the context of usual care are allowed to continue. After the 32-week follow-up, the participants in the UC group have the option to follow a modified version of the AET or CBT interventions without supervision.

Participants will be given the option to undergo a quantitative muscle MRI of the upper legs. The MRI is additional and not mandatory to participate in the study. The investigators will include a maximum of 10 participants per group. Participants will undergo the MRI twice: before intervention at baseline and after intervention at 20 weeks follow-up.

Furthermore, a qualitative study will be conducted to explore the experiences of participants in both the AET and CBT groups. Semi-structured interviews, based on a topic list, will be held with 10 participants from each intervention group separately. These interviews will take place within three months after the intervention phase has ended.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. A clinical diagnosis of myasthenia gravis (ocular or generalized) as defined by the Dutch national guideline (category "definite" or "probable" MG).
3. The diagnosis of MG was made at least a year ago and the MG is stable, as determined by the treating neurologist.
4. Patients who use the following medication: prednisone, intravenous immunoglobulin (IVIg), complement inhibitor (e.g. Eculizumab), neonatal Fc receptor (FcRn) inhibitor (e.g. Efgartigimod) have been on a stable dosing regimen for at least one month.
5. MGFA Clinical Classification of disease severity I-IV.
6. Clinically relevant fatigue (a score ≥ 27 on the CIS-fatigue).
7. Ability to walk and exercise.
8. Ability to understand the requirements of the study and provide written informed consent.

Exclusion Criteria:

1. The patient is unable to fill out the study questionnaires or be interviewed in Dutch, or is unable to undergo the tests needed for the study, or is unable to give informed consent for participation in the study.
2. The patient is unable to use the activity tracker and digital infrastructure provided.
3. Co-morbidity interfering with AET or affecting exercise response and exercise capacity, including severe cardiopulmonary co-morbidity, as assessed by the investigator.
4. Co-morbidity interfering with CBT, a clinical diagnosis of depression or a score ≥12 on the Hospital Anxiety and Depression Scale (HADS) depression subscale, as assessed by the investigator.
5. Use of beta blockers.
6. The patient is already engaged in strenuous exercise more than twice a week.
7. The patient is already undergoing cognitive behavioural therapy.
8. Pregnancy or intention to become pregnant during the study.

Exclusion Criterion for muscle MRI 1. Inability to undergo MRI.

- In case of uncertainty about the MRI-contraindications, the MR-safety commission of the Radiology department will decide whether this subject can be included in the study or not.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
A change in CIS-fatigue in the AET and CBT group, compared to UC, before and after intervention. | Assessed after 4 weeks and 20 weeks.
  Fatigue measured on the Checklist Individual Strength (CIS-) fatigue subscale. The CIS-fatigue consists of eight questions on fatigue experienced during the previous two weeks. Each question is scored on a 7-point Likert scale and a score ≥ 27 indicates increased fatigue and a score ≥ 35 indicates severe fatigue. A higher score means more severe fatigue. A decline of ≥8 is considered clinically relevant. The total score of the fatigue subscale ranges from 8-56 (the total score of the CIS questionnaire ranges from 20-140).

SECONDARY OUTCOMES:
A change in CIS-fatigue in the AET group compared to the CBT group before and after intervention and during follow-up. | Assessed after 20 weeks and 32 weeks.
  Fatigue measured on the Checklist Individual Strength (CIS-) fatigue subscale. The CIS-fatigue consists of eight questions on fatigue experienced during the previous two weeks. Each question is scored on a 7-point Likert scale and a score ≥ 35 indicates severe fatigue. A higher score means more severe fatigue. A decline of ≥8 is considered clinically relevant. The total score of the fatigue subscale ranges from 8-56 (the total score of the CIS questionnaire ranges from 20-140).
A sustained change in CIS-fatigue after AET or CBT intervention at 32 weeks (12 weeks post-intervention). | Assessed after 32 weeks.
  Fatigue measured on the Checklist Individual Strength (CIS-) fatigue subscale. The CIS-fatigue consists of eight questions on fatigue experienced during the previous two weeks. Each question is scored on a 7-point Likert scale and a score ≥ 35 indicates severe fatigue. A higher score means more severe fatigue. A decline of ≥8 is considered clinically relevant. The total score of the fatigue subscale ranges from 8-56 (the total score of the CIS questionnaire ranges from 20-140).
A long term change in CIS-fatigue after AET or CBT intervention at 52 weeks. | Assessed after 52 weeks.
  Fatigue measured on the Checklist Individual Strength (CIS-) fatigue subscale. The CIS-fatigue consists of eight questions on fatigue experienced during the previous two weeks. Each question is scored on a 7-point Likert scale and a score ≥ 35 indicates severe fatigue. A higher score means more severe fatigue. A decline of ≥8 is considered clinically relevant. The total score of the fatigue subscale ranges from 8-56 (the total score of the CIS questionnaire ranges from 20-140).
The number of completed AET or CBT sessions to investigate participants' compliance with a 16 week AET or CBT program. | Assessed after 20 weeks.
  Compliance with the AET program: at least 40 sessions (of a total of 48 sessions).
  Compliance with the CBT program: at least 8 sessions.
A change in the use of MG medication before and after AET or CBT intervention, compared to usual care. | Assessed after 20 weeks and 32 weeks.
  Changes in types of medication and changes in dosages of medication.
A change in MG Quality of Life 15-item (MG-QoL 15r) Scale after AET or CBT intervention compared to usual care. | Assessed after 4 weeks, 20 weeks, 32 weeks and 52 weeks.
  MG-QoL 15r consists of 15 items with a total score of 0-30; a higher score indicating worse health-related quality of life.
A clinically relevant change in MG Activities of Daily Living (MG-ADL) Scale after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
  MG-ADL consists of 8 items with a total score of 0-24; a higher score indicating more severe disease. ≥2 points change is considered a clinically relevant change.
A clinically relevant change in Quantitative MG (QMG) Scale after AET or CBT intervention compared to usual care | Assessed after 4 weeks and 20 weeks.
  QMG consists of 13 items with a total score of 0-39; a higher score indicating more severe disease. ≥3 points change is considered a clinically relevant change.
Changes in amount of weekly vigorous intensity physical activity, as measured by the number of minutes per week that the heart rate reaches at least 70% of maximum heart rate after AET or CBT intervention compared to usual care. | Assessed after 4 weeks, 20 weeks, 32 weeks and 52 weeks.
  Measured by a remote activity tracker.
A change in cardiorespiratory fitness (CRF) after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
  Measured by an aerobic fitness test (Steep Ramp Test (SRT)) measuring the Wpeak.
A change in CIS-activity after AET or CBT intervention compared to usual care. | Assessed after 4 weeks, 20 weeks, 32 weeks and 52 weeks.
  Checklist Individual Strength (CIS-) activity subscale is a subscale consisting of 3 questions with each question scored on a 7-point Likert scale with a total score of 3-21; a higher score indicating less activity. This subscale is not validated for use as standalone outcome measure in MG and does not have an established cut-off score or threshold for clinical relevance
A change in International Physical Activity Questionnaire - Short Form (IPAQ-SF) after AET or CBT intervention compared to usual care. | Assessed on day 1, after 4 weeks and 20 weeks.
  IPAQ-SF consists of 7 questions; a higher score indicating more strenuous activity.
A change in CIS-concentration and -motivation after AET or CBT intervention compared to usual care. | Assessed after 4 weeks, 20 weeks, 32 weeks and 52 weeks.
  Checklist Individual Strength (CIS-) concentration and motivation subscales are subscales consisting of 5 and 4 questions respectively with each question scored on a 7-point Likert scale; a higher score indicating more concentration problems or lower motivation respectively. These subscales are not validated for use as standalone outcome measures in MG and do not have an established cut-off scores or thresholds for clinical relevance.
A change in Hospital Anxiety and Depression Scale (HADS) after AET or CBT intervention compared to usual care. | Assessed on day 1, after 4 weeks and 20 weeks.
  HADS consists of 14 items divided into two subscales with each question scored on a 4-point Likert scale; a higher score indicating more symptoms. The total score per subscale (anxiety, depression) ranges from 0-21.
A change in Visual Analogue Scale (VAS-pain) after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
  VAS-pain is a continuous scale with a total score of 0-10; a higher score indicating greater pain intensity.
A change in Pittsburgh Sleep Quality Index (PSQI) after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
  PSQI consists of 19 items with a total score of 0-21; a higher score indicating worse sleep quality.
A change in the social interaction subscale of the Sickness Impact Profile (SIP) after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
  SIP consists of 136 items that cover 12 health categories. The social interaction category consists of 20 items; a higher score indicating more health-related behavioural problems. The total score of the SIP ranges from 0-100.
A change in EQ-5D-5L after AET or CBT intervention compared to usual care. | Assessed on day 1, after 4 weeks, 20 weeks, 32 weeks and 52 weeks.
  The 5-level EQ-5D (EQ-5D-5L) version consists of 25 questions divided into 5 domains and a continuous scale.
Changes in the relation of fatigue with CRP serum levels at baseline and after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
Changes in the relation of fatigue with AChR antibody serum levels at baseline and after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
Changes in the relation of fatigue with MuSK antibody serum levels at baseline and after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
Changes in the relation of fatigue with muscle MRI parameters at baseline and after AET or CBT intervention compared to usual care. | Assessed after 4 weeks and 20 weeks.
  M. rectus femoris and m. biceps femoris caput longe: fat fraction, cross sectional area (mm2), contractile cross sectional area (mm2), T2 relaxation time (ms), fractional anisotropy (FA) and mean diffusivity (MD).
  Optional for up to 10 participants per group.
To record participants' subjective perspectives to qualitatively assess the process and outcome of a 16 week AET or CBT program. | Within 3 months after the intervention phase.
  Semi-structured interviews to get insight into the experiences of patients regarding the process of the interventions, interpretation of effects, and explore factors which influence the implementation of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn R. Tannemaat, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No